CLINICAL TRIAL: NCT01735773
Title: The Relationship of Prohepcidin Levels With Anemia and Inflammatory Markers in Non-diabetic Uremic Patients: A Controlled Study
Brief Title: Role of Prohepcidin in Uremic Patients
Status: Completed | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HEPCIDIN-HASEKI
Record Dates: First submitted 2012-11-26; First posted 2012-11-28 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Inflammation; Chronic Kidney Disease
Keywords: hemodialysis; inflammation; iron; peritoneal dialysis; prohepcidin; uremia
MeSH Terms: conditions — Inflammation; Renal Insufficiency, Chronic; Uremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Hemodialysis group: Patients on chronic hemodialysis program
- Peritoneal dialysis group: Patients on chronic peritoneal dialysis program
- Pre-dialysis group: Patients with chronic kidney disease stage-4
- Control group: Healthy volunteers

SUMMARY:
The investigators aimed to study the effect of prohepcidin levels on hematologic parameters and inflammatory markers in non-diabetic uremic patients. The investigators selected three groups of patients: Hemodialysis group, peritoneal dialysis group and the group with stage 4 chronic kidney disease. A control group was formed from healthy volunteers also. Each group has been planned to be formed of about 25 patients. Diabetic patients were excluded. Prohepcidin, hsCRP, IL-6, fibrinogen have been planned to be studied besides other routine biochemical analysis including hematological ones.

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis and peritoneal dialysis patients who had been on dialysis therapy for more than 3 months,
* age between 18-80 years,
* patients with creatinine clearance between 15-30 ml/min.

Exclusion Criteria:

* age less than 18 or more than 80,
* diabetic patients,
* current active infectious or inflammatory disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We selected three groups of patients: Hemodialysis group, peritoneal dialysis group and the group with stage 4 chronic kidney disease. A control group was formed from healthy volunteers also.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
prohepcidin level | Six months
  Prohepcidin levels will be compared with other inflammatory markers.

SECONDARY OUTCOMES:
Anemia and inflammatory markers | Six months
  Correlations of prohepcidin levels with anemia and inflamatory markers

CONTACTS AND LOCATIONS:
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Turkey (Türkiye)